CLINICAL TRIAL: NCT00061698
Title: CBT vs CBT Plus Parent Training for Girls With Depression
Brief Title: Treatment for Depressed Preadolescent Girls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH063998 (NIH); R01MH063998 (NIH); DSIR 84-CTS
Record Dates: First submitted 2003-06-03; First posted 2003-06-04 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Behavior Therapy Child Only (Active Comparator): Participants completed 20 sessions of CBT
  Interventions: Behavioral: Cognitive Behavior Therapy Child Only
- CBT plus Parent training (Active Comparator): Child participants completed 20 sessions of CBT and parents completed 8 sessions of parent training
  Interventions: Behavioral: Cognitive Behavior Therapy Child Only; Behavioral: CBT plus Parent Training
- Minimal Contact Control (No Intervention): Participants waited 12 weeks for treatment but their safety and well-being were monitored during this time

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy Child Only — Participants learned and applied coping skills, problem solving, cognitive restructuring strategies and built a positive core belief.
  Arms: CBT plus Parent training; Cognitive Behavior Therapy Child Only
Behavioral: CBT plus Parent Training — Participants learned and applied coping skills, problem solving, cognitive restructuring strategies and built a positive core belief. Parents learned skills that helped their child to apply the strategies they learned. Parents learned how to better communicate positive information that helped their child build a positive core belief. Parents learned how to use reinforcement to support healthy behavior.
  Arms: CBT plus Parent training

SUMMARY:
This study will compare the effectiveness of three therapies for the treatment of depression in preadolescent girls.

DETAILED DESCRIPTION:
Depressive disorders during childhood are virulent, long-lasting disorders that are a risk factor for the development of future depressive episodes and other psychiatric difficulties. A dysfunctional family environment is a possible pathway to the development of depression in adolescents. The family environment is an especially salient context for the development of depression in preadolescent girls.

Depression is expressed differently between male and female adolescents; girls may not benefit as much as boys from treatments such as cognitive behavioral therapy (CBT) because the treatments may not target disturbances and skills that are specific to preadolescent girls. This study will identify effective treatments for depression in preadolescent girls.

Depressed participants are randomly assigned to receive CBT, CBT plus parent training (PT), or a minimal contact control (MCC). The CBT group receives treatment twice a week for 10 weeks. Participants in the CBT plus PT group receive therapy sessions and group treatment for 10 weeks. Participants in the MCC group meet with a research associate once a week for 10 weeks. During the control visits, the child's depressive symptoms are assessed, but no advice or treatment is given. Participants are assessed at baseline, post-treatment, and at yearly follow-up visits for up to 4 years. School performance, home environment, and the impact of the interventions on parent adjustment are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Depressive Disorder

Exclusion Criteria:

* Learning disability or limited intellectual ability
* Health-related illness that would prevent the patient from completing the research study

Ages: 9 Years to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2002-04; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

REFERENCES:
- [Background] Cole DA, Cai L, Martin NC, Findling RL, Youngstrom EA, Garber J, Curry JF, Hyde JS, Essex MJ, Compas BE, Goodyer IM, Rohde P, Stark KD, Slattery MJ, Forehand R. Structure and measurement of depression in youths: applying item response theory to clinical data. Psychol Assess. 2011 Dec;23(4):819-33. doi: 10.1037/a0023518. Epub 2011 May 2. PMID 21534696
- [Background] Stark, K. D. (2008). Experiences Implementing the ACTION Treatment Program: Implications for Preventive Interventions. Clinical Psychology: Science and Practice, 15, 342 - 345.
- [Background] Stapleton LM, Sander JB, Stark KD. Psychometric properties of the Beck Depression Inventory for Youth in a sample of girls. Psychol Assess. 2007 Jun;19(2):230-5. doi: 10.1037/1040-3590.19.2.230. PMID 17563204
- [Result] Morey, M. E., Arora, P., & Stark, K. D. (in press). Multiple-Stage Screening of Youth Depression in Schools. Psychology in the Schools.